CLINICAL TRIAL: NCT03332017
Title: An International, Phase 2, Open-Label, Randomized Study of BGB-3111 Combined With Obinutuzumab Compared With Obinutuzumab Monotherapy in Relapsed/ Refractory Follicular Lymphoma
Brief Title: A Study Comparing Obinutuzumab and BGB-3111 Versus Obinutuzumab Alone in Treating R/R Follicular Lymphoma
Acronym: ROSEWOOD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-212; 2017-001552-54 (EudraCT Number); CTR20220712 (Other: ChinaDrugTrials)
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Relapsed/Refractory Follicular Non-Hodgkin Lymphoma
Keywords: Relapsed/Refractory Follicular non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — zanubrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obinutuzumab (Experimental): Obinutuzumab 1000 milligrams (mg) intravenously on Days 1, 8, and 15 of Cycle 1; Day 1 of Cycles 2 to 6; and then every 8 weeks until unacceptable toxicity, withdrawal of consent, loss of clinical benefit, or disease progression; each cycle is 28 days
  Interventions: Drug: Obinutuzumab
- Zanubrutinib + Obinutuzumab (Experimental): Zanubrutinib 160 mg twice a day orally with or without food; Obinutuzumab 1000 mg intravenously on Days 1, 8, and 15 of Cycle 1; Day 1 of Cycles 2 to 6; and then every 8 weeks until unacceptable toxicity, withdrawal of consent, loss of clinical benefit, or disease progression; each cycle is 28 days
  Interventions: Drug: Zanubrutinib; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Zanubrutinib — Oral administration as a capsule
  Other Names: BGB-3111; Brukinsa
  Arms: Zanubrutinib + Obinutuzumab
Drug: Obinutuzumab — Intravenous administration
  Other Names: Gazyva

SUMMARY:
he purpose of the study is to evaluate the efficacy, safety, and tolerability BGB-3111 plus obinutuzumab versus obinutuzumab alone in participants with relapsed/refractory non-Hodgkin follicular lymphoma.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed diagnosis of B-cell follicular lymphoma
2. ≥2 prior systemic treatments for follicular lymphoma.
3. Previously received an anti-CD20 antibody and an appropriate alkylator-based combination therapy.
4. Disease progression after completion of most recent therapy or refractory disease.
5. Presence of measurable disease.
6. Availability of archival tissue confirming diagnosis.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2.
8. Adequate renal and hepatic function.

Key Exclusion Criteria:

1. Prior exposure to a Bruton's tyrosine kinase (BTK) inhibitor.
2. Known central nervous system involvement by leukemia or lymphoma.
3. Evidence of transformation from follicular lymphoma to other aggressive histology.
4. Allogeneic hematopoietic stem cell transplantation within 12 months of enrollment
5. Prior malignancy within the past 2 years, except for curatively treated basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix of breast, or localized Gleason score 6 prostate cancer.
6. Clinically significant cardiovascular disease.
7. Major surgery ≤ 4 weeks prior to start of study treatment.
8. Active fungal, bacterial or viral infection requiring systemic treatment.
9. History of severe bleeding disorder.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2024-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (89):
- United States (4):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University of Illinois At Chicago, Chicago, Illinois
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Duke University, Durham, North Carolina
- Australia (12):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Saint Vincents Hospital Sydney, Darlinghurst, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Icon Cancer Centre Wesley, Auchenflower, Queensland
  - Icon Cancer Foundation, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Peninsula Private Hospital, Frankston, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Belarus (3):
  - Minsk City Clinical Oncological Dispensary, Minsk
  - Nn Alexandrov National Cancer Centre of Belarus, Minsk
  - Vitebsk Regional Clinical Oncology Dispensary, Vitebsk
- Bulgaria (4):
  - University Multiprofile Hospital For Active Treatment Dr Georgi Stranski, Pleven
  - Acibadem City Clinic Mhat Tokuda Ead, Sofia
  - University Multiprofile Hospital For Active Treatment Saint Ivan Rilski, Sofia
  - University Multiprofile Hospital For Active Treatment Alexandrovska, Sofia
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec
- China (12):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- Czechia (4):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Slezska Nemocnice V Opave, Opava
  - Vseobecna Fakultni Nemocnice V Praze, Prague
- France (9):
  - Centre Hospitalier Universitaire Damiens Hopital Sud, Amiens
  - Centre de Lutte Contre Le Cancer Institut Bergonie, Bordeaux
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Clinique Louis Pasteur, Esseylesnancy
  - Necker University Hospital, Paris
  - Chu Bordeaux Hopital Haut Leveque, Pessac
  - Chu Hopital Lyon Sud, PierreBenite
  - Centre Hospitalier Universitaire de Poitier Hopital de La Miletrie Hopital Jean Bernard, Poitiers
  - Centre Henri Becquerel, Rouen
- Klinikum Augsburg, Ii Medizinische Klinik, Augsburg, Germany
- Italy (7):
  - Azienda Ospedaliera Policlinico Di Bari, Bari
  - Policlinico Sorsola Malpighi, Aou Di Bologna, Bologna
  - Ospedale San Raffaele, Milan
  - Istituto Europeo Di Oncologia, Milan
  - Azienda Ospedaliero Universitaria Di Parma, Parma
  - Unita Di Ematologia, Dipartimento Di Ematologia Ed Oncologia, Ravenna
  - Ospedale Di Circolo E Fondazione Macchi, Varese
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Aotearoa Clinical Trials, Auckland
  - Christchurch Hospital, Christchurch
- Poland (4):
  - Malopolskie Centrum Medyczne Sc, Krakow
  - Wielospecjalistyczne Centrum Onkologii I Traumatologii Im M Kopernika W Lodzi, Lodz
  - Centrum Onkologii Ziemi Lubelskiej, Lublin
  - Szpital Wojewodzki W Opolu, Opole
- Russia (4):
  - State Healthcare Institution Oncologic Dispensary No Health Department of Krasnodar Region, Sochi, Krasnodarskiy Kray
  - N N Blokhin Russian Cancer Research Center Konstantin Laktionov, Moscow, Moscow
  - Central City Hospital, Yekaterinburg, Sverdlovsk Oblast
  - Tula Area Clinical Hospital, Tula, Tula Oblast
- South Korea (4):
  - Kyungpook National University Hospital, Daegu, Daegu Gwang'yeogsi
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, Seoul, Seoul Teugbyeolsi
- Spain (8):
  - Institut Catala Doncologia, Barcelona
  - Hospital Universitario Puerta Del Mar, Cadiz
  - Md Anderson Cancer Center Madrid Spain, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario de Salamanca, Salamanca
- Taiwan (4):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital West Campus, Taipei
- United Kingdom (4):
  - The Royal Bournemouth and Christchurch Hospitals Nhs Foundation, Bournemouth
  - The Leeds Teaching Hospitals Nhs Trust, Leeds
  - Barts Health Nhs Trust, London
  - Norfolk and Norwich University Hospitals Nhs Foundation Trust, Norwich

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Trotman J, Folwer N, Auer R, Flowers C, Reed W, Stern JC, Huang J, Zinzani PL. Phase 2 Obinutuzumab Zanubrutinib (BGB-3111) in Patients with Relapsed/Refractory Follicular Lymphoma (R/R FL). American Society of Clinical Oncology, 2018.
- [Background] Fowler N, Trotman J, Auer R, Flowers C, Reed W, Marimpietri C, Huang J, Zinzani PL.Randomized phase 2 zanubrutinib (BGB-3111) + obinutuzumab (obi) vs obi monotherapy in patients (pts) with relapsed/refractory follicular lymphoma (R/R FL). American Society of Clinical Oncology. 2019
- [Background] Fowler NH, Trotman J, Auer R, Flowers CR, Reed WF, Ivanova E, Huang J, Zinzani PL.Randomized Phase 2 Zanubrutinib (BGB-3111) + Obinutuzumab vs Obinutuzumab Monotherapy in Patients with Relapsed/Refractory Follicular Lymphoma (R/R FL). American Society of Hematology. 2019
- [Derived] Trotman J, Zinzani PL, Song Y, Delarue R, Kim P, Ivanova E, Korde R, Mayer J, De Oliveira AC, Assouline SE, Flowers CR, Barnes G. Patient-reported outcomes in patients with relapsed or refractory follicular lymphoma treated with zanubrutinib plus obinutuzumab versus obinutuzumab monotherapy: results from the ROSEWOOD trial. Curr Med Res Opin. 2024 Nov;40(11):1863-1871. doi: 10.1080/03007995.2024.2409837. Epub 2024 Oct 14. PMID 39376156
- [Derived] Zinzani PL, Mayer J, Flowers CR, Bijou F, De Oliveira AC, Song Y, Zhang Q, Merli M, Bouabdallah K, Ganly P, Zhang H, Johnson R, Martin Garcia-Sancho A, Provencio Pulla M, Trneny M, Yuen S, Tilly H, Kingsley E, Tumyan G, Assouline SE, Auer R, Ivanova E, Kim P, Huang S, Delarue R, Trotman J. ROSEWOOD: A Phase II Randomized Study of Zanubrutinib Plus Obinutuzumab Versus Obinutuzumab Monotherapy in Patients With Relapsed or Refractory Follicular Lymphoma. J Clin Oncol. 2023 Nov 20;41(33):5107-5117. doi: 10.1200/JCO.23.00775. Epub 2023 Jul 28. PMID 37506346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in multiple study centers in Australia, Europe, China, Taiwan, South Korea, and North America. Data are presented as of the primary completion data cut-off date of 08OCT2021.
Groups:
- Zanubrutinib + Obinutuzumab: Zanubrutinib 160 milligrams (mg) twice a day orally with or without food; Obinutuzumab 1000 mg intravenously on Days 1, 8, and 15 of Cycle 1; Day 1 of Cycles 2 to 6; and then every 8 weeks until unacceptable toxicity, withdrawal of consent, loss of clinical benefit, or disease progression; each cycle is 28 days
Period: Overall Study
Arm/Group | Obinutuzumab | Zanubrutinib + Obinutuzumab
Started | 72 | 145
Completed | 0 | 0
Not Completed | 72 | 145
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 17 | 16
Not completed — Withdrawal by Subject | 6 | 14
Not completed — Other | 1 | 3
Not completed — Remained in Study (Ongoing) | 47 | 110

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) analysis set includes all randomized participants. Data are presented as of the primary completion data cut-off date of 08OCT2021.
Groups:
- Obinutuzumab: Obinutuzumab 1000 mg intravenously on Days 1, 8, and 15 of Cycle 1; Day 1 of Cycles 2 to 6; and then every 8 weeks until unacceptable toxicity, withdrawal of consent, loss of clinical benefit, or disease progression; each cycle is 28 days
- Total: Total of all reporting groups
Arm/Group | Obinutuzumab | Zanubrutinib + Obinutuzumab | Total
Number analyzed (Participants) | 72 | 145 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (12.81) | 61.1 (11.98) | 61.7 (12.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 70 | 109
  Male | 33 | 75 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 63 | 131 | 194
  Unknown or Not Reported | 7 | 10 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 51 | 106 | 157
  Asian | 17 | 31 | 48
  Not Reported | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) by Independent Review Committee (IRC) Assessment
Description: ORR is defined as the percentage of participants who achieve either complete response (CR) or partial response (PR) as best overall response, as assessed by the IRC using Lugano Classification for Non-Hodgkin Lymphoma
Time Frame: Through primary analysis data cut-off date of 08OCT2021 (up to approximately 3 years and 11 months)
Population: Intent-To-Treat (ITT) analysis set includes all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab | Zanubrutinib + Obinutuzumab
Number analyzed (Participants) | 72 | 145
percentage of participants | 45.8 [34.0 to 58.0] | 68.3 [60.0 to 75.7]
Statistical Analysis 1: Comparison: Obinutuzumab vs Zanubrutinib + Obinutuzumab; Test type: Superiority; p = 0.0017, Cochran-Mantel-Haenszel; P-value was stratified by rituximab-refractory status, number of prior lines of therapy, and geographic region per interactive response technology

2. Secondary Outcome: Overall Response Rate (ORR) as Assessed by the Investigator
Time Frame: Up to approximately 7 years
Reporting Status: Not Posted

3. Secondary Outcome: Duration of Response (DOR)
Time Frame: Up to approximately 7 years
Reporting Status: Not Posted

4. Secondary Outcome: Progression Free Survival (PFS)
Time Frame: Up to approximately 7 years
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival (OS)
Time Frame: Up to approximately 7 years
Reporting Status: Not Posted

6. Secondary Outcome: Complete Response Rate
Time Frame: Up to approximately 7 years
Reporting Status: Not Posted

7. Secondary Outcome: Complete Metabolic Response Rate
Time Frame: Up to approximately 7 years
Reporting Status: Not Posted

8. Secondary Outcome: Time to Response (TTR)
Time Frame: Up to approximately 7 years
Reporting Status: Not Posted

9. Secondary Outcome: Health-Related Quality of Life (HRQOL) as Assessed by The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Time Frame: Up to approximately 7 years
Reporting Status: Not Posted

10. Secondary Outcome: Health-Related Quality of Life (HRQOL) as Assessed by The 5-level EQ-5D Version (EQ-5D-5L)
Time Frame: Up to approximately 7 years
Reporting Status: Not Posted

11. Secondary Outcome: Occurrence and Severity of Treatment-emergent Adverse Events (TEAEs)
Description: Safety and Tolerability
Time Frame: Up to approximately 7 years
Reporting Status: Not Posted

12. Secondary Outcome: Apparent Clearance (CL/F) of Zanubrutinib
Time Frame: Day 1 Cycle 1 and Day 2 Cycle 2: Predose
Reporting Status: Not Posted

13. Secondary Outcome: Area Under the Curve From 0 to 12 Hours Post Dose (AUC0-12)
Time Frame: Day 1 Cycle 1 and Day 2 Cycle 2: Pre-dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the first dose up to 30 days after the last dose of zanubrutinib or 90 days after the last dose of obinutuzumab; through primary analysis data cut-off date of 08OCT2021 (up to approximately 3 years and 11 months)
Description: All-cause mortality is reported for all randomized participants. Serious and other adverse events includes all randomized participants who received ≥ 1 dose of any study treatment .
Arm/Group | Obinutuzumab | Zanubrutinib + Obinutuzumab
All-Cause Mortality (participants affected / at risk) | 17/72 | 16/145
Serious Adverse Events (participants affected / at risk) | 19/71 | 45/143
Other Adverse Events (participants affected / at risk) | 57/71 | 121/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obinutuzumab (N=71) | Zanubrutinib + Obinutuzumab (N=143)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Necrotic lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spigelian hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Swelling face (General disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (2) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (3) | 1 (2)
COVID-19 pneumonia (Infections and infestations) | 2 (3) | 4 (5)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Myelitis (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 7 (9)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (2) | 1 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Vascular access site infection (Infections and infestations) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (4)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obinutuzumab (N=71) | Zanubrutinib + Obinutuzumab (N=143)
Anaemia (Blood and lymphatic system disorders) | 6 (10) | 13 (42)
Neutropenia (Blood and lymphatic system disorders) | 11 (21) | 16 (47)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (19) | 26 (76)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 10 (12)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 6 (6)
Constipation (Gastrointestinal disorders) | 5 (5) | 19 (23)
Diarrhoea (Gastrointestinal disorders) | 12 (14) | 23 (35)
Nausea (Gastrointestinal disorders) | 8 (11) | 12 (16)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 7 (9)
Vomiting (Gastrointestinal disorders) | 4 (7) | 9 (14)
Asthenia (General disorders) | 6 (8) | 13 (18)
Chills (General disorders) | 4 (6) | 3 (4)
Fatigue (General disorders) | 8 (10) | 20 (24)
Oedema peripheral (General disorders) | 3 (4) | 3 (3)
Peripheral swelling (General disorders) | 4 (4) | 2 (3)
Pyrexia (General disorders) | 12 (16) | 16 (25)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1)
Conjunctivitis (Infections and infestations) | 3 (3) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 8 (10)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 9 (12)
Pneumonia (Infections and infestations) | 3 (3) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 9 (11)
Urinary tract infection (Infections and infestations) | 3 (3) | 10 (13)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 10 (11)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 7 (7)
Infusion related reaction (Injury, poisoning and procedural complications) | 7 (10) | 4 (4)
Neutrophil count decreased (Investigations) | 7 (18) | 23 (61)
Platelet count decreased (Investigations) | 10 (26) | 24 (67)
White blood cell count decreased (Investigations) | 2 (5) | 13 (49)
Decreased appetite (Metabolism and nutrition disorders) | 4 (6) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (5) | 8 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 13 (15)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 2 (4) | 6 (6)
Post herpetic neuralgia (Nervous system disorders) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 17 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 14 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (12)
Erythema (Skin and subcutaneous tissue disorders) | 3 (5) | 4 (5)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 10 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (10) | 10 (11)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (8)
Haematoma (Vascular disorders) | 1 (1) | 5 (5)
Hypertension (Vascular disorders) | 3 (4) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03332017/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT03332017/SAP_001.pdf